CLINICAL TRIAL: NCT03593265
Title: Calculation of Normal MUNIX Variation in an Healthy Population
Brief Title: MUNIX Variability in Healthy Subjects
Acronym: MUNIX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-45
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy group (Experimental): healthy subjects MUNIX will be performed
  Interventions: Other: MUNIX

INTERVENTIONS:
Other: MUNIX — Motor unit number index in 4 muscles: tibialis anterior, abductor digiti mini, abductor pollicis brevis et deltoideus

SUMMARY:
Motor unit number index (MUNIX) is an electrophysiological technique that estimates the number of motor units in a muscle. This data can be changed by natural evolution or by treatment in peripheral neuropathy. Alfortunately, normal value for MUNIX variation does not exist. Thus, it is difficult to assume improvement or worsening of the MUNIX for an individual subject.

Our objective is to calculate normal variation of MUNIX in 4 muscles : tibialis anterior, abductor digiti mini, abductor pollicis brevis et deltoideus. Measurement will be performed at inclusion and 3 monthes later in 100 healthy subjects. This trial will be prospective in several French centres sepecialized in neuromuscular evaluation

DETAILED DESCRIPTION:
Motor unit number index (MUNIX) is an electrophysiological technique that estimates the number of motor units in a muscle. This data can be changed by natural evolution or by treatment in peripheral neuropathy. Alfortunately, normal value for MUNIX variation does not exist. Thus, it is difficult to assume improvement or worsening of the MUNIX for an individual subject.

Our objective is to calculate normal variation of MUNIX in 4 muscles: tibialis anterior, abductor digiti mini, abductor pollicis brevis et deltoideus. Measurement will be performed at inclusion and 3 monthes later in 100 healthy subjects. This trial will be prospective in several French centres sepecialized in neuromuscular evaluation

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without neuromuscular disoreders or others diseases which can interfer with MUNIX measurement
* More than 18 years old

Exclusion Criteria:

* Less than 18 years old
* Diseases which can interfer with MUNIX measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
MUNIX | 3 months
  motor unit number inedx in 4 muscles: tibialis anterior, abductor digiti mini, abductor pollicis brevis et deltoideus

SECONDARY OUTCOMES:
MUSIX | 3 months
  muscle size index
CMAP amplitudes | 3 months
  the greatest possible amplitude

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France